CLINICAL TRIAL: NCT04588493
Title: Human Adjuvant Disease as a Cause of Secondary Lower Extremity Lymphedema
Brief Title: Secondary Lymphedema Due to Human Adjuvant Disease
Status: Completed | Type: Observational
Sponsor: Hospital Angeles del Pedregal (Other)
Responsible Party: Principal Investigator, javier lopez, Principal investigator, Plastic and reconstructive surgeon staff, MBA, FACS, Hospital Angeles del Pedregal
Other Study IDs: HAD and lymphedema
Record Dates: First submitted 2020-10-08; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Lymphedema, Secondary; Lymphedema of Leg; Granuloma, Foreign-Body
Keywords: human adjuvant disease
MeSH Terms: conditions — Lymphedema; Neoplasm Metastasis; Granuloma, Foreign-Body

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lower extremity Lymphoscintigraphy — Study of lymphoscintigraphy (LCG) abnormalities in a group of patients with history of infiltration of modeling substances in buttocks and hips and complain about lower extremities edema. LCG was performed and evaluated by a single nuclear medicine specialist through injection of the sulfur nanocolloid Technetium 99m, injected intradermal and interdigital in bilateral toes. Dynamic studies were requested for all patients. Standardized acquisition times at 15, 30, 60 and 120 minutes after injection were taken. The following parameters were considered to obtain the transport index in each pelvic limb: transport kinematics, distribution pattern, index time for the appearance of regional lymph nodes, number and collection of colloids in lymph nodes and presence and quality of the colloid uptake by the lymphatic vessels. Summation of these five components resulted in the transport index, which could range from 0 to 45 points

SUMMARY:
This observational, descriptive, retrospective study the clinical and imaging findings of 10 lower legs of 5 patients with previous history of injection of modeling substances for cosmetic purposes at buttocks and hips ande developed lower limb edema. Lower limb lymphedema index and lymphoscintigraphy findings were evaluated and reported.

DETAILED DESCRIPTION:
Lymphoscintigraphy findings were reported with the Transport index (TI), were any value over 5 will represent abnormalities in lymphatic function.

ELIGIBILITY:
Inclusion Criteria:

* Both sex
* Over 18 years old
* History of injection of modelling substances for cosmetic purposes
* History of lower limb edema

Exclusion Criteria:

* History of primary lower limb lymphedema
* Reject to participate
* Confirmed other causes of edema

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with history of injection of modeling substances for cosmetic purposes (non Federal Drug Administration-approved substances) in buttocks and presenting lower limb edema
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Transport Index | 4 months
  Transport index in each pelvic limb: transport kinematics, distribution pattern, index time for the appearance of regional lymph nodes, number and collection of colloids in lymph nodes and presence and quality of the colloid uptake by the lymphatic vessels. Summation of these five components resulted in the transport index, which could range from 0 to 45 points; less than 5 means a normal study, higher scores represent abnormal or pathological results

SECONDARY OUTCOMES:
Lower extremity lymphedema index | 4 months
  For Lower extremity lymphedema (LEL) index we first added up cross-sectional areas of the extremities in 5 parts where circumferences were measured, making an approximation that the cross-sections are perfect circles. We made use of the sum of the cross-sectional area's property of being proportional to the sum of the square of the circumference to simplify the calculation of the formula. Finally, we divided the number by BMI to make corrections for the body type, and the obtained value was defined as the LEL index. Dividing the sum by BMI corrected the index according to the body type. LEL index < 250 corresponded to LEL stage I, 250 to 300 corresponded to LEL stage II, 300 to 350 corresponded to LEL stage III, and > 350 corresponded to LEL stage IV

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Angeles Pedregal, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Study will be published and we will share the results of transport index and lower limb lymphedema index. Also the standardized method to acquire the lymphoscintigraphic evaluation.
Supporting Information: Study Protocol, CSR